CLINICAL TRIAL: NCT00137150
Title: Comparison of Outcome and Complications Encountered in Flapless Surgery and Immediate Loading Versus the Classical Surgical Approach and Loading After 6-8 Weeks in the Posterior Maxilla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Institut Straumann AG (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004/420
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Placement of implants

SUMMARY:
This study is a comparison of outcome and complications encountered in flapless surgery and immediate loading versus the classical surgical approach and loading after 6-8 weeks in the posterior maxilla.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older

Exclusion Criteria:

* Smoking
* Medical risk patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2005-01; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Implant survival at 6-12 months

SECONDARY OUTCOMES:
Prosthetic complications
Patient opinion

CONTACTS AND LOCATIONS:
Overall Officials: Hugo De Bruyn, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be